CLINICAL TRIAL: NCT05424692
Title: Vitro 3D Drug Sensitivity Detection of Micro Tumor (PTC) Combined with Tumor Whole Exon (WES) Sequencing Technology to Guide Postoperative Adjuvant Treatment Strategy and Prognosis of Colorectal Cancer
Brief Title: Drug Sensitivity Detection of Micro Tumor (PTC) to Guide Postoperative Adjuvant Treatment Strategy of Colorectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PekingUMCHPTC
Record Dates: First submitted 2022-05-03; First posted 2022-06-21 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-09

CONDITIONS: Colon Cancer; Rectal Cancer; Chemotherapy Effect; PTC; Exon Mutation
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Formyltetrahydrofolates; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PTC test group (Experimental): The adjuvant chemotherapy scheme was selected according to the 3D drug sensitivity test results of micro tumor (PTC) in vitro
  Interventions: Drug: 5-fluorouracil + formyltetrahydrofolate/Oxaliplatin + 5-fluorouracil + formyltetrahydrofolate/Irinotecan + 5-fluorouracil + formyltetrahydrofolate/Cetuximab + 5-fluorouracil + formyltetrahydrofolate
- control group (No Intervention): Making adjuvant chemotherapy strategy based on clinical experience

INTERVENTIONS:
Drug: 5-fluorouracil + formyltetrahydrofolate/Oxaliplatin + 5-fluorouracil + formyltetrahydrofolate/Irinotecan + 5-fluorouracil + formyltetrahydrofolate/Cetuximab + 5-fluorouracil + formyltetrahydrofolate — Choose chemotherapeutic drugs（5-fluorouracil + formyltetrahydrofolate/Oxaliplatin + 5-fluorouracil + formyltetrahydrofolate/Irinotecan + 5-fluorouracil + formyltetrahydrofolate/Cetuximab + 5-fluorouracil + formyltetrahydrofolate） based on PTC drug sensitivity results.
  Other Names: PTC drug sensitivity results
  Arms: PTC test group

SUMMARY:
The research objectives is to compare vitro 3D drug sensitivity test results of micro tumor (PTC) with the clinical outcomes of patients, evaluate the consistency between the test results of the technology platform and the clinical prognosis, and explore the decision-making value and guiding significance of this technology in assisting the precise treatment of colorectal cancer. The completion of this study will provide real-world data support for the clinical application of micro tumor (PTC) in vitro 3D drug sensitivity detection technology, and provide more valuable reference basis for realizing the individualization and accuracy of colorectal cancer treatment and improving the clinical benefit rate.

DETAILED DESCRIPTION:
The study is a multi agency prospective cohort study in China. The subjects were patients aged 18 ~ 75 years with colorectal cancer diagnosed by histopathology or cytology. They must be colorectal cancer patients who have at least one assessable tumor focus, need adjuvant therapy after radical surgery, and have not received neoadjuvant therapy， ECoG physical condition score ≤ 2 points. And they must be voluntarily participate in and sign informed consent.

The patients were randomly divided into PTC drug sensitivity test group and control group. The PTC drug sensitivity test group selected the adjuvant chemotherapy scheme according to the 3D drug sensitivity test results of micro tumor (PTC) in vitro. The control group made adjuvant chemotherapy strategy according to clinical experience. All exon (WES) data collection was used to predict postoperative survival in both groups.

The primary endpoint was the non inferiority test, and the 3-year disease-free survival rate was T-C >- Δ

ELIGIBILITY:
Inclusion Criteria:

* Age 18 ~ 75 years old, regardless of gender
* Patients with colorectal cancer diagnosed by histopathology or cytology
* Colorectal cancer patients who need adjuvant therapy after radical surgery and have not received neoadjuvant therapy
* Having at least one assessable tumor focus
* ECoG physical condition score ≤ 2 points
* Voluntarily participate and sign informed consent

Exclusion Criteria:

* Patients diagnosed with metastasis
* Patients who cannot obtain tumor samples
* Pregnant and lactating women
* Patients with poor compliance
* Patients with severe cardiovascular and cerebrovascular complications who cannot receive adjuvant treatment
* Patients with other malignant tumors
* Suffering from serious mental and nervous system diseases
* The researchers believe that patients should not be selected for this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
The difference of 3-year disease-free survival rate of patients in both group | 3 years
  Follow-up the survival status of patients, and calculate 3-year disease-free survival rate of patients in both group

SECONDARY OUTCOMES:
The relation between TMB and clinical outcomes | 3 years
  Use tumor whole exon (WES) sequencing to detect the Tumor Mutation Burden (TMB) of patients, and use correlation analysis to detect whether it's risk factor of clinical outcomes.
The relation between MSI and clinical outcomes | 3 years
  Use tumor whole exon (WES) sequencing to detect the Microsatellite Instability (MSI) of patients, and use correlation analysis to detect whether it's risk factor of clinical outcomes.
The relation between dMMR and clinical outcomes | 3 years
  Use tumor whole exon (WES) sequencing to detect the Deficient Mismatch Repair (dMMR) of patients, and use correlation analysis to detect whether it's risk factor of clinical outcomes.
The difference of clinical outcomes of patients in both group | 3 years
  Follow-up the health status and weather tumor recurrence and metastasis of patients, and evaluate whether the test results of extended drug regimen correspond with clinical outcomes
The difference of TTP of patients in both group | 3 years
  Follow-up the results of patients' periodic reviews and calculate Time To Progress (TTP） of patients in both group, and use survival analysis to detect whether the two group has difference in TTP.
The difference of ORR of patients in both group | three years
  Follow-up the results of patients' periodic reviews and calculate Objective Response Rate (ORR） of patients in both group, and use survival analysis to detect whether the two group has difference in ORR.
The difference of DFS of patients in both group | 3 years
  Follow-up the results of patients' periodic reviews and calculate Disease Free Survival (DFS) of patients in both group, and use survival analysis to detect whether the two group has difference in DFS.
The difference of PFS of patients in both group | 3 years
  Follow-up the results of patients' periodic reviews and calculate Progress Free Survival (PFS） of patients in both group, and use survival analysis to detect whether the two group has difference in PFS.
The difference of OS of patients in both group | 3 years
  Follow-up the results of patients' periodic reviews and calculate Overall Survival (OS） of patients in both group, and use survival analysis to detect whether the two group has difference in OS.

CONTACTS AND LOCATIONS:
Overall Officials: Guole Lin, Study Chair — Peking Union Medical College Hospital; Jiaolin Zhou, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Gramont A, Figer A, Seymour M, Homerin M, Hmissi A, Cassidy J, Boni C, Cortes-Funes H, Cervantes A, Freyer G, Papamichael D, Le Bail N, Louvet C, Hendler D, de Braud F, Wilson C, Morvan F, Bonetti A. Leucovorin and fluorouracil with or without oxaliplatin as first-line treatment in advanced colorectal cancer. J Clin Oncol. 2000 Aug;18(16):2938-47. doi: 10.1200/JCO.2000.18.16.2938. PMID 10944126
- [Background] Siegel R, DeSantis C, Virgo K, Stein K, Mariotto A, Smith T, Cooper D, Gansler T, Lerro C, Fedewa S, Lin C, Leach C, Cannady RS, Cho H, Scoppa S, Hachey M, Kirch R, Jemal A, Ward E. Cancer treatment and survivorship statistics, 2012. CA Cancer J Clin. 2012 Jul-Aug;62(4):220-41. doi: 10.3322/caac.21149. Epub 2012 Jun 14. PMID 22700443
- [Background] Goldberg RM, Sargent DJ, Morton RF, Fuchs CS, Ramanathan RK, Williamson SK, Findlay BP, Pitot HC, Alberts SR. A randomized controlled trial of fluorouracil plus leucovorin, irinotecan, and oxaliplatin combinations in patients with previously untreated metastatic colorectal cancer. J Clin Oncol. 2004 Jan 1;22(1):23-30. doi: 10.1200/JCO.2004.09.046. Epub 2003 Dec 9. PMID 14665611
- [Background] Yin S, Xi R, Wu A, Wang S, Li Y, Wang C, Tang L, Xia Y, Yang D, Li J, Ye B, Yu Y, Wang J, Zhang H, Ren F, Zhang Y, Shen D, Wang L, Ying X, Li Z, Bu Z, Ji X, Gao X, Jia Y, Jia Z, Li N, Li Z, Ji JF, Xi JJ. Patient-derived tumor-like cell clusters for drug testing in cancer therapy. Sci Transl Med. 2020 Jun 24;12(549):eaaz1723. doi: 10.1126/scitranslmed.aaz1723. PMID 32581131
- [Background] Cassidy J, Clarke S, Diaz-Rubio E, Scheithauer W, Figer A, Wong R, Koski S, Lichinitser M, Yang TS, Rivera F, Couture F, Sirzen F, Saltz L. Randomized phase III study of capecitabine plus oxaliplatin compared with fluorouracil/folinic acid plus oxaliplatin as first-line therapy for metastatic colorectal cancer. J Clin Oncol. 2008 Apr 20;26(12):2006-12. doi: 10.1200/JCO.2007.14.9898. PMID 18421053
- [Background] Gao H, Korn JM, Ferretti S, Monahan JE, Wang Y, Singh M, Zhang C, Schnell C, Yang G, Zhang Y, Balbin OA, Barbe S, Cai H, Casey F, Chatterjee S, Chiang DY, Chuai S, Cogan SM, Collins SD, Dammassa E, Ebel N, Embry M, Green J, Kauffmann A, Kowal C, Leary RJ, Lehar J, Liang Y, Loo A, Lorenzana E, Robert McDonald E 3rd, McLaughlin ME, Merkin J, Meyer R, Naylor TL, Patawaran M, Reddy A, Roelli C, Ruddy DA, Salangsang F, Santacroce F, Singh AP, Tang Y, Tinetto W, Tobler S, Velazquez R, Venkatesan K, Von Arx F, Wang HQ, Wang Z, Wiesmann M, Wyss D, Xu F, Bitter H, Atadja P, Lees E, Hofmann F, Li E, Keen N, Cozens R, Jensen MR, Pryer NK, Williams JA, Sellers WR. High-throughput screening using patient-derived tumor xenografts to predict clinical trial drug response. Nat Med. 2015 Nov;21(11):1318-25. doi: 10.1038/nm.3954. Epub 2015 Oct 19. PMID 26479923
- [Derived] Qiu X, Li R, Xie G, Ning N, Wang Z, Zhou J, Liu G, Tang Q, He Z, Yang L, Lu J, Li P, Lin G. In vitro 3D drug sensitivity testing for patient-derived tumor-like cell clusters and whole-exome sequencing to personalize postoperative treatment: A study protocol for a multicenter randomized controlled trial. PLoS One. 2025 Jul 14;20(7):e0326760. doi: 10.1371/journal.pone.0326760. eCollection 2025. PMID 40658653